CLINICAL TRIAL: NCT05786950
Title: Neural Respiratory Drive of Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YLS2020(172)
Record Dates: First submitted 2023-03-04; First posted 2023-03-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: neural respiratory drive; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Intervention Model Description: the responds of the neural respiratory drive of the chronic obstructive pulmonary disease patients after inhaling bronchodilator(3mg salbutamol and 500μg ipratropium, Boehringer Ingelheim Limited, Germany).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bronchodilators (Experimental): compound ipratropium bromide solution (3mg salbutamol and 500μg ipratropium, Boehringer Ingelheim Limited, Germany)
  Interventions: Drug: compound ipratropium bromide solution (3mg salbutamol and 500μg ipratropium, Boehringer Ingelheim Limited, Germany)

INTERVENTIONS:
Drug: compound ipratropium bromide solution (3mg salbutamol and 500μg ipratropium, Boehringer Ingelheim Limited, Germany) — inhaled compound ipratropium bromide solution (3mg salbutamol and 500μg ipratropium, Boehringer Ingelheim Limited, Germany)

SUMMARY:
To investigate the relationship among the neural respiratory drive (NRD), the sensation of the dyspnea and the effect of the bronchodilator on each stage COPD patients.

DETAILED DESCRIPTION:
Different stage COPD subjects were recruited. Administration of bronchodilators was prohibited 24 hours prior to the experiment. After the application of topical anesthesia (10% xylocaine) the subject was asked to swallow the multipair esophageal electrode catheter through the nose into their right position. At the first period, the stable signals of spontaneous breathing (about 10 minutes) were collected as the baseline data. At the second period, each subject inhaled compound ipratropium bromide solution (3mg salbutamol and 500μg ipratropium, Boehringer Ingelheim Limited, Germany). A multi-pair esophageal electrode catheter with 10 coils that provided five pairs of electrodes was used to obtain the NRD signals. All NRD signals the were recorded before and after the compound ipratropium bromide solution was inhaled (about 10 minutes). The subjects scored their comfort sensation with a visual analog scale (VAS) ranging from 0 (best) to 10 (worst) at each period.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of COPD was made according to the global initiative for chronic obstructive lung disease (GOLD) guideline.

-

Exclusion Criteria:

(1) Malignancy （2）Severe cardiovascular diseases （3）Neuromuscular and chest wall deformity (4) Cardiovascular instability (hypotension, arrhythmias, myocardial infarction) (5) Change in mental status; uncooperative patients (6) Extreme obesity （7）renal failure and severe blood electrolyte disturbances (8) Asthma-

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
the change of the neural respiratory drive | 20 minutes
  the change of the neural respiratory drive

SECONDARY OUTCOMES:
comfort sensation | 20 minutes
  The subjects scored their comfort sensation with a visual analog scale (VAS) ranging from 0 (best) to 10 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: jianheng zhang, MD, Principal Investigator — State Key Laboratory of Respiratory Disease
Locations (1):
- 1State Key Laboratory of Respiratory Disease, National clinical research center for respiratory disease, Guangzhou Institute of respiratory health. 2The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided